CLINICAL TRIAL: NCT01903499
Title: Satiety Effects of Beef Compared to Beans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 1212E25808
Record Dates: First submitted 2013-02-20; First posted 2013-07-19 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bean patty (Active Comparator): Bean Patty
  Interventions: Other: Other: Bean patty; Other: Other: Beef patty
- Beef patty (Active Comparator): Beef patty
  Interventions: Other: Other: Bean patty; Other: Other: Beef patty

INTERVENTIONS:
Other: Other: Bean patty
Other: Other: Beef patty

SUMMARY:
The satiety effects of beef will be compared to beans. Beef is hypothesized to be more satiating than beans.

DETAILED DESCRIPTION:
Subjects will consume 2 different meatloaf lunches and satiety will be measured by visual analogue scales. They will consume an ad lib snack after 3 hours and food intake will be measured.

ELIGIBILITY:
Inclusion Criteria:

healthy, non-smoking, BMI of 18-27, non-dieting, typically consumes breakfast/lunch

Exclusion Criteria:

distaste for beans, vegetarian, current smoker, restrained eating habits, recent weight change, history of significant disease of past medical history, pregnant, lactating irregular menstrual cycle

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
satiety | 180 minutes
  Measure satiety by visual analogue scale (VAS)

SECONDARY OUTCOMES:
food intake | 180 minutes
  assorted snacks provided to assess food intake variation between treatments

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States